CLINICAL TRIAL: NCT03536325
Title: A Double-blind, Placebo-controlled, Randomized, Single Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Guselkumab Following a Single Intravenous Administration in Healthy Japanese Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Guselkumab Following a Single Intravenous Administration in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108478; CNTO1959CRD1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2018-05-15; First posted 2018-05-24 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Healthy
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: Guselkumab Dose 1 or Placebo (Experimental): Participants will receive Dose 1 of guselkumab or matching placebo as an intravenous (IV) infusion on Day 1.
  Interventions: Drug: Guselkumab Dose 1; Drug: Placebo
- Cohort 2: Guselkumab Dose 2 or Placebo (Experimental): Participants will receive Dose 2 of guselkumab or matching placebo as an IV infusion on Day 1.
  Interventions: Drug: Guselkumab Dose 2; Drug: Placebo
- Cohort 3: Guselkumab Dose 3 or Placebo (Experimental): Participants will receive Dose 3 of guselkumab or matching placebo as an IV infusion on Day 1 based on safety data results received from Cohort 1 and 2.
  Interventions: Drug: Guselkumab Dose 3; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab Dose 1 — Participants will receive Dose 1 of guselkumab on Day 1.
  Other Names: CNTO1959
  Arms: Cohort 1: Guselkumab Dose 1 or Placebo
Drug: Guselkumab Dose 2 — Participants will receive Dose 2 of guselkumab on Day 1.
  Other Names: CNTO1959
  Arms: Cohort 2: Guselkumab Dose 2 or Placebo
Drug: Guselkumab Dose 3 — Participants will receive Dose 3 of guselkumab on Day 1.
  Other Names: CNTO1959
  Arms: Cohort 3: Guselkumab Dose 3 or Placebo
Drug: Placebo — Participants will receive matching placebo on Day 1.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of guselkumab following single-dose intravenous (IV) infusion in Japanese healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy with no clinically significant abnormalities as determined by medical history, physical examination, blood chemistry assessments, hematologic assessments, urinalysis, measurement of vital signs, and electrocardiogram (ECG)
* Must agree to use an adequate contraception method as deemed appropriate by the investigator; to always use a condom during intercourse and to not donate sperm during the study and for 16 weeks after study drug administration
* Must be a nonsmoker or agree to smoke no more than 10 cigarettes or 2 cigars per day throughout the study, if the inpatient site allows. However, if smoking is not allowed in the inpatient site, smokers will not be allowed to smoke while inpatient cannot use nicotine replacement products during the inpatient period, but may smoke at other times during the study, up to the maximum stated above
* Must agree to abstain from alcohol intake 48 hours before study drug administration and during the inpatient period of the study. After this time, participants must not consume more than 10 grams of alcohol per day for the duration of the study

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, gastro-intestinal disease, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Has had major surgery, (for example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study
* Has known allergies, hypersensitivity, or intolerance to guselkumab or its excipients
* Any medical contraindications preventing study participation

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to approximately 20 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Day 1: predose, end of infusion (EOI) and 8 hours (h) post dose; Day 2: 24 h post dose; Day 3: 48 h post dose; Day 4: 72 h post dose; Day 5: 96 h; Day 6: 120 h; Day 7: 144 h post dose; Days 15, 22, 29, 43, 57, 71, 85, 99, and 113
  The Cmax is the maximum observed serum concentration.
Area Under the Serum Concentration Versus Time Curve from Time 0 to the Time Corresponding to the Last Quantifiable Plasma Concentration (AUC[0-last]) | Day 1: predose, EOI and 8 h post dose; Day 2: 24 h post dose; Day 3: 48 h post dose; Day 4: 72 h post dose; Day 5: 96 h; Day 6: 120 h; Day 7: 144 h post dose; Days 15, 22, 29, 43, 57, 71, 85, 99, and 113
  The AUC(0-last) is the area under the serum concentration-time curve from time 0 to last quantifiable concentration.
Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Day 1: predose, EOI and 8 h post dose; Day 2: 24 h post dose; Day 3: 48 h post dose; Day 4: 72 h post dose; Day 5: 96 h; Day 6: 120 h; Day 7: 144 h post dose; Days 15, 22, 29, 43, 57, 71, 85, 99, and 113
  The AUC(0-infinity) is the area under the serum concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the serum concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Terminal half-life (t1/2) | Day 1: predose, EOI and 8 h post dose; Day 2: 24 h post dose; Day 3: 48 h post dose; Day 4: 72 h post dose; Day 5: 96 h; Day 6: 120 h; Day 7: 144 h post dose; Days 15, 22, 29, 43, 57, 71, 85, 99, and 113
  Terminal half-life (t1/2) is the time measured for the serum concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Systemic Clearance (CL) | Day 1: predose, EOI and 8 h post dose; Day 2: 24 h post dose; Day 3: 48 h post dose; Day 4: 72 h post dose; Day 5: 96 h; Day 6: 120 h; Day 7: 144 h post dose; Days 15, 22, 29, 43, 57, 71, 85, 99, and 113
  CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose is estimated by dividing the total administered dose by the plasma Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]).
Volume of Distribution (Vz) | Day 1: predose, EOI and 8 h post dose; Day 2: 24 h post dose; Day 3: 48 h post dose; Day 4: 72 h post dose; Day 5: 96 h; Day 6: 120 h; Day 7: 144 h post dose; Days 15, 22, 29, 43, 57, 71, 85, 99, and 113
  The Vz is total volume of distribution at terminal phase after IV administration, defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Number of Participants with Antibodies to Guselkumab | Day 1: predose; and Days 15, 29, 57, and 113
  Number of participants with antibodies to guselkumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Japan